CLINICAL TRIAL: NCT06566092
Title: A Phase 1, Multicenter, Open-label, 2-stage, Single-arm Study to Evaluate the Safety and Tolerability of an Autologous Tumor-infiltrating Lymphocytes (TIL) Regimen and Preliminary Antitumor Activity of TIL in Pediatric, Adolescent, and Young Adult Participants With Relapsed or Refractory Solid Tumors
Brief Title: Study of Autologous Tumor-Infiltrating Lymphocytes in Pediatric, Adolescent, and Young Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-PED-101
Record Dates: First submitted 2024-07-17; First posted 2024-08-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Soft Tissue Sarcoma; Primary Central Nervous System Carcinoma; Melanoma; Rhabdomyosarcoma; Ewing Sarcoma
Keywords: Tumor Infiltrating Lymphocytes; TIL; Pediatric; Soft Tissue Sarcoma; Primary Nervous System Carcinoma; PCNS; Rhabdomyosarcoma; RMS; Ewing Sarcoma; EWS
MeSH Terms: conditions — Sarcoma; Melanoma; Rhabdomyosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Intervention Model Description: Participants are assigned one of three arms depending on their tumor type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rhabdomyosarcoma (RMS) (Experimental)
  Interventions: Biological: LN-145/LN-144
- Ewing Sarcoma (EWS) (Experimental)
  Interventions: Biological: LN-145/LN-144
- Primary Central Nervous System Tumor (Experimental)
  Interventions: Biological: LN-145/LN-144
- Melanoma (Experimental)
  Interventions: Biological: LN-145/LN-144

INTERVENTIONS:
Biological: LN-145/LN-144 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes.

SUMMARY:
This study is planned to test the safety and tolerability of the TIL regimen. The study will also test how well TIL fights cancer. The study will enroll children, teenagers, and young adults with solid tumors that have returned or are not responding to treatment for whom no effective standard-of-care treatment options exist.

Study details include:

* The study will last up to 2 years after the TIL infusion (Day 0) for each person.
* The treatment will last up to 10 days for each person.
* Study visits will be every 2 weeks until Day 42, every 6 weeks until Month 6, and every 3 months until Year 2.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 8 kg and ≤ 21 years of age at the time of informed consent and assent.
2. Histologically or cytologically confirmed recurrent or refractory solid tumor (Rhabdomyosarcoma, Ewing sarcoma, primary CNS malignancies, melanoma) after standard therapy which has failed all available curative therapy.
3. Acceptable performance status and an estimated life expectancy of > 6 months.
4. At least one resectable lesion (solitary or aggregate lesions) for TIL generation.
5. Following tumor resection for TIL generation, the participant will have at least one remaining measurable lesion for response assessment.
6. Preplanned surgical procedure(s) will take place at least 14 days (for major operative procedures) prior to the tumor resection.
7. All prior anticancer treatment-related AEs should be recovered, exceptions are peripheral neuropathy, alopecia, vitiligo, or medically controlled endocrine dysfunction.
8. Agreement to abide by the protocol indicated contraception use, including refraining from donating sperm or eggs (ova, oocytes), as appropriate for the age and sexual activity of pediatric, adolescent, and young adult participants and as required by local regulations.
9. Signed informed consent and assent when applicable.
10. Written authorization for use and disclosure of protected health information.
11. Ability to adhere to the study visit schedule and other protocol requirements.
12. Acceptable hematologic parameters.
13. Adequate organ function.
14. Modified Ross criteria class 1 and an LVFS > 25% or an LVEF ≥ 50%.
15. Adequate pulmonary function.
16. Participant and/or the legal guardian who provided consent is willing for the participant to receive optimal supportive care.
17. A legal guardian or primary caregiver must be available to help the study-site personnel ensure follow-up and accompany the participant to the study site on each assessment day according to the SoA.

Exclusion Criteria:

1. Participant with a non-CNS tumor has symptomatic untreated brain metastases and/or carcinomatous meningitis.
2. Participant has an active or uncontrolled intercurrent illness(es) that would pose increased risks for study participation.
3. Participants are not eligible if they experience uncontrolled seizures.
4. Participants with history of intracranial hemorrhage/spinal cord hemorrhage.
5. Participant has active uveitis that requires active treatment.
6. Participant has significant psychiatric disease or substance abuse in the investigator's opinion that would prevent adequate informed consent.
7. Participant has any form of primary or acquired immunodeficiency.
8. History of clinically significant chronic obstructive pulmonary disease, asthma, interstitial lung disease, or other chronic lung disease.
9. History of hypersensitivity reaction to any components of the study intervention.
10. Any other condition that in the investigator's judgment would significantly increase the risks of participation.
11. Any complication or delayed healing from an excisional procedure that in the investigator's opinion would increase the risks of participation.
12. Another primary malignancy within the previous 3 years.
13. History of allogeneic cell or organ transplant.
14. Requiring systemic steroid therapy higher than the physiologic replacement dose.
15. Received or will receive a live or attenuated vaccination within 28 days prior to the start of the NMA-LD.
16. Any active viral, bacterial, or fungal infection requiring ongoing systemic treatment.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Treatment-Emergent Adverse Events | Up to 24 months
  To evaluate the safety and tolerability of the TIL regimen that occurs from the start of TIL infusion and up to 30 days after TIL infusion per CTCAE.

SECONDARY OUTCOMES:
Objective Response Rate | Up to 24 months
  To evaluate the proportion of participants who have confirmed complete response (CR) or partial response (PR) per RECIST v1.1 or RAPNO.
Duration of Response | Up to 24 months
  To measure the time that criteria are met for complete response (CR) or partial response (PR) per RECIST v1.1 or RAPNO.
Disease Control Rate | Up to 24 months
  To measure by the percentage of participants with best overall confirmed response of complete response (CR) or partial response (PR) at any time or stable disease (SD) for at least 4 weeks per RECIST v1.1 or RAPNO.
Progression-Free Survival | Up to 24 months
  To evaluate the time from the date of the TIL infusion until disease progression per RECIST v1.1 or RAPNO.
Overall Survival | Up to 24 months
  To measure the time from the date of TIL infusion to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Study Team, Study Director — Iovance Biotherapeutics
Locations (5):
- United States (5):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York